CLINICAL TRIAL: NCT05050747
Title: An Open-label Prospective Controlled Study to Assess the Effect of Intrauterine Adminstration of HCG Versus Endometrial Injury by Pipelle on the Ongoing Pregnancy Rate in Patients with Unexplained Infertility Undergoing Ovulation Induction
Brief Title: Study to Assess the Effect of Intrauterine Adminstration of HCG Versus Endometrial Injury by Pipelle
Status: Completed | Type: Observational
Sponsor: Wael Elbanna Clinic (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Wael Elbanna, Managing director for Wael Elbanna Clinic, Wael Elbanna Clinic
Other Study IDs: Elbanna_002
Record Dates: First submitted 2021-08-13; First posted 2021-09-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2021-09

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Arm 1: Women with unexplained infertility undergoing ovulation induction following intrauterine adminstration of HCG on the day of trigger
  Interventions: Drug: HCG is introduced at day of trigger intra-uterine
- Arm 2: Women with unexplained infertility undergoing ovulation induction following endometrial injury by pipelle on day 8-9 of the same cycle of ovulation induction
  Interventions: Device: endometrial injury by pipelle
- Arm 3: Women with unexplained infertility undergoing ovulation induction following intrauterine adminstration of placebo on the day of trigger

INTERVENTIONS:
Drug: HCG is introduced at day of trigger intra-uterine — hcg is introduced
  Groups: Arm 1
Device: endometrial injury by pipelle — endometrial injury using pipelle on day 8-9 on the same cycle of ovulation
  Groups: Arm 2

SUMMARY:
Our study aims to describe the effect of the intrauterine adminstration of HCG versus the endometrial injury by pipelle on the ongoing pregnancy rate and the biochemical pregnancy rate in women with unexplained infertility undergoing ovulation induction. Also to describe the effect on the first trimester miscarriage rate, ectopic pregnancy rate, and multiple pregnancy.This study is an open-label, prospective, controlled study, multi-center study.

The study participants' relevant medical records will be collected and reviewed after obtaining informed consent for the participants. The study materials that will be used will include blood tests, and ultrasound. The study will involve three study arms.

DETAILED DESCRIPTION:
Our study aims to describe the effect of the intrauterine adminstration of HCG versus the endometrial injury by pipelle on the ongoing pregnancy rate and the biochemical pregnancy rate in women with unexplained infertility undergoing ovulation induction. Also to describe the effect on the first trimester miscarriage rate, ectopic pregnancy rate, and multiple pregnancy.This study is an open-label, prospective, controlled study, multi-center study.

The study participants' relevant medical records will be collected and reviewed after obtaining informed consent for the participants. The study materials that will be used will include blood tests, and ultrasound. The study will involve three study arms:

Arm 1: Women with unexplained infertility undergoing ovulation induction following intrauterine adminstration of HCG on the day of trigger Arm 2: Women with unexplained infertility undergoing ovulation induction following endometrial injury by pipelle on day 8-9 of the same cycle of ovulation induction Arm 3: Women with unexplained infertility undergoing ovulation induction following intrauterine adminstration of placebo on the day of trigger

Primary and secondary key measurements will be used in the study.

The primary measures will include:

* Signs of ongoing pregnancy Presence of intrauterine gestational sac at 12 weeks Presence of fetal heart pulsation at 12 weeks
* Two serum β-HCG levels in 48hrs interval to emphasis biochemical pregnancy

The secondary key measures will include:

* Occurance of abortion in the 1st trimester
* Appearance of ectopic pregnancy diagnosis by:

Ultrasound Serum β-HCG level Symptoms of pain and bleeding

* Signs of multiple pregnancy Number of intrauterine gestational sacs Number of fetal poles Number of fetal heart pulsations
* Recording the the baseline characteristics of the study participants

ELIGIBILITY:
Inclusion Criteria:

1. Women with primary or secondary infertility due to unexplained infertility
2. The age group of these women was 25-35 years
3. BMI 18.5-29.9 kg/m2
4. Normal hormone profile (FSH <10 mIU/ml on day 2-3 and AMH more than 1)
5. Euthyroid state or controlled thyroid state
6. Bilateral free spill on HSG

Exclusion Criteria:

1. Patients with severe male factor infertility; serum analysis count < 10 million sperms /mL - sperm motility<15% - 96%<abnormal morphology)
2. Stage III or IV endometriosis
3. Bilateral tubal factor infertility
4. Premature ovarian failure
5. Polycystic ovary syndrome
6. Uterine cavity abnormality
7. Recurrent spontaneous abortion

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will include women with unexplained infertility undergoing ovulation induction following either:
  1. Intrauterine adminstration of HCG
  2. Endometrial injury by pipelle
  3. Intrauterine adminstration of placebo
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Signs of ongoing pregnancy | Till the end of the 1st trimester
  Recording the following for the three arms of the study:
  * Signs of ongoing pregnancy Presence of intrauterine gestational sac at 12 weeks Presence of fetal heart pulsation at 12 weeks
  * Two serum β-HCG levels in 48hrs interval to emphasis biochemical pregnancy

SECONDARY OUTCOMES:
occurance of abortion or ectopic or multiple pregnancy | Till the end of the 1st trimester
  Recording the following for the three arms of the study:
  * Occurance of abortion in the 1st trimester
  * Appearance of ectopic pregnancy diagnosis by:
  Ultrasound Serum β-HCG level Symptoms of pain and bleeding
  - Signs of multiple pregnancy Number of intrauterine gestational sacs Number of fetal poles Number of fetal heart pulsations
Recording the baseline characteristics of the study participants | Before study intervention
  age , height , weight , body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Wael Elbanna Clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided